CLINICAL TRIAL: NCT03821597
Title: The Effect of Intraoperative Sequential Compression Devices on Fibrinolysis in Plastic Surgery Outpatients: A Randomized Trial
Brief Title: Sequential Compression Devices Effect on Fibrinolysis in Plastic Surgery Outpatients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swanson Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Swanson 010
Record Dates: First submitted 2019-01-27; First posted 2019-01-30 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Blood Coagulation Disorder
Keywords: Fibrinolysis, sequential compression devices
MeSH Terms: conditions — Blood Coagulation Disorders

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, controlled study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequential compression devices (Experimental): Sequential compression devices (SCDs) are applied during surgery.
  Interventions: Procedure: Sequential compression devices (SCDs)
- No sequential compression devices (Active Comparator): No sequential compression devices are applied.
  Interventions: Procedure: No sequential compression.

INTERVENTIONS:
Procedure: Sequential compression devices (SCDs) — Application of sequential compression devices in surgery.
  Arms: Sequential compression devices
Procedure: No sequential compression. — No sequential compression devices are applied.
  Arms: No sequential compression devices

SUMMARY:
This study investigates a possible fibrinolytic effect of sequential compression devices (SCDs). These devices have been used for decades to reduce risk of deep venous thrombosis (DVT). However, a randomized study in plastic surgery outpatients has not been done. This study is undertaken to remedy that deficiency in our knowledge base.

DETAILED DESCRIPTION:
Protocol: The Effect of Intraoperative Sequential Compression Devices on Fibrinolysis in Plastic Surgery Outpatients

1. Study Synopsis

   Deep venous thrombosis (DVT) is a serious and potentially life-threatening surgical complication. Sequential compression devices (SCDs), also called intermittent pneumatic compression, are widely used by surgeons in an effort to reduce risk. In addition to a possible mechanical effect, some investigators believe that these devices reduce the coagulability of blood by altering the fibrinolytic balance. This investigation is meant to evaluate any possible effect of these devices on fibrinolytic activity.

   The SCDs are not being investigated for a new indication. This study is meant to determine whether these commonly used devices have any effect on blood coagulability. This study is not intended to determine whether SCDs affect DVT rates.
2. Background

   The investigator (ES) has conducted a literature search on this topic. There is no published prospective randomized study available investigating a possible fibrinolytic effect of SCDs in surgical patients. Therefore any clinical benefit remains speculative.
3. Objective

   The use of this device is well-recognized. The rationale for using SCDs in this study is to investigate their potential effect on blood coagulability.
4. Subject Selection

   The proposed study is a prospective randomized study involving 50 consecutive plastic surgery outpatients who consent to participate. Twenty-five patients will have sequential compression devices applied and 25 patients will not be treated with these devices and will serve as controls. All subjects are adults aged 18 or over undergoing elective cosmetic surgery, including both men and women.

   All patients, men and women, are included with no exclusion criteria (that go beyond exclusion criteria for elective outpatient surgery). Pregnant women are not surgical candidates and are excluded (women in the reproductive age group are routinely checked with a pregnancy test). There are no contraindications to SCDs among patients undergoing elective outpatient plastic surgery. Patients with coagulopathies that would represent a contraindication for surgery, or significant diseases (heart disease, uncontrolled diabetes) are excluded. Oral contraceptive use is permitted.

   The purpose of including patients who are not treated with SCDs is to have a control group, which is mandatory in a randomized study. The sample size of 50 was obtained from an a priori power analysis and sample size calculation to allow statistical significance at an alpha value of 0.05. The use of SCDs is not a standard of care requirement. Their efficacy remains controversial, with no high-level (i.e. Level 1) support.

   All patients receive measures to reduce the risk of DVT. No muscle relaxation is used during surgery to preserve the calf muscle pump. Patients ambulate immediately after surgery. In addition, patients are monitored with ultrasound surveillance to ensure the early detection and treatment of any DVTs that may develop postoperatively. Patients do not normally receive anti-platelet therapy because of the increased risk of bleeding.

   Patients with contraindications to the use of SCDs will be excluded from the study. These conditions include suspected active or untreated DVT, pulmonary edema, congestive heart failure, thrombophlebitis or an active infection, vein ligation, gangrene, dermatitis, open wounds, a recent skin graft, massive edema or extreme deformity of the leg, neuropathy, legs that are insensitive to pain, or when increased venous or lymphatic return is undesirable. None of these conditions is present in healthy patients undergoing elective cosmetic surgery, which form the study group.
5. Study Procedures

   The duration of the study is 2 months, sufficient to obtain data for 50 consecutive patients. All patients are plastic surgery outpatients undergoing elective cosmetic procedures. The consent discussion will take place between the principal investigator and the patient. All surgery will be performed by the study author at a state-licensed ambulatory surgery center, the Surgery Center of Leawood, KS.

   Patients already have IV access at the time of surgery. A blood sample (2 cc) will be drawn immediately before surgery and at 1-hour intervals during surgery and in the recovery room. The blood samples will be analyzed at an outside laboratory for tissue plasminogen activator (tPA) and plasminogen activator inhibitor-1 (PAI-1) levels at these time points. The number of blood draws will be determined by the length of the operation and time in the recovery room. The last blood sample is taken at the hourly interval that immediately precedes the patient's discharge from the recovery room.

   All patients will undergo ultrasound surveillance. This diagnostic test is painless, noninvasive, and highly accurate for detecting DVTs. Scans are performed before surgery, on the day after surgery, and 1 week after surgery.
6. Risk/Safety Information

   There is no risk or discomfort to the patient and the amount of blood drawn is minuscule. There added risks associated with SCD sleeves are very rare, such as skin irritation, nerve compression, and patient falls, although the latter problem is impossible because the devices are removed prior to the patient waking up from surgery.
7. Monitoring/Reporting of Adverse Events

   Any adverse event will be monitored by the principal investigator and reported to patients, although none is expected. The principal investigator will collect, assess, and follow-up on any adverse events. Any adverse events will be reported, including to the Institutional Review Board (IRB) and regulatory authorities.
8. Study Oversight

   There are no foreseeable circumstances that would abort the study. The study and data will be available for auditing.

   Data Management
9. Data will be analyzed by a biostatistician.
10. IRB Review/Ethics Informed Consent

    This study meets the standard of equipoise in that there is no known benefit of SCDs in preventing DVTs in plastic surgery outpatients. SCDs harmlessly compress the calves and are known to be extremely safe. Each subject will receive full and adequate verbal and written information. Consenting patients will read and sign the Informed Consent document prior to taking part in the study and prior to surgery. Any change in the protocol will be submitted for review. This study is undertaken in accordance with ethical principles that have their origin in the Declaration of Helsinki and are consistent with Good Clinical Practice and applicable regulatory requirements. This study will be conducted in accordance with the regulations of the U.S. Food and Drug Administration (FDA) applicable laws and IRB requirement.
11. Confidentiality

    Pooled data will be evaluated without any identifying information by a Ph.D. biostatistician. There is no opportunity for violation of patient privacy. Blood samples will only include a number (Patient 1, patient 2, etc.) and the date and time of the blood draw with no patient identifying information sent to the lab (Quest Laboratories). Patient information is kept within a secure location within the office of the principal investigator in accordance with HIPAA requirements. No patient identification will accompany any publications of the study. The data are open to inspection by any regulatory authorities.
12. Intended Use of the Data

The data will be evaluated to determine whether or not the null hypothesis is confirmed (i.e. whether SCDs affect blood coagulability). It is expected that the study findings will be published in the medical literature.

Disclosure

The author has no financial interest in any of the products, devices, or drugs used in this study. The author has no conflicts of interest to disclose. The investigator has no financial interest in ultrasound or the device used. There is no outside funding for this study.

ELIGIBILITY:
Inclusion Criteria:

* All healthy patients aged 18 or more.

Exclusion Criteria:

* These conditions include suspected active or untreated DVT, pulmonary edema, congestive heart failure, thrombophlebitis or an active infection, vein ligation, gangrene, dermatitis, open wounds, a recent skin graft, massive edema or extreme deformity of the leg, neuropathy, legs that are insensitive to pain, or when increased venous or lymphatic return is undesirable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-01-27 (Actual)

PRIMARY OUTCOMES:
Change in plasma levels of tissue plasminogen activator and plasminogen activator inhibitor-1 | 1-2 months
  Laboratory testing of serum levels

CONTACTS AND LOCATIONS:
Overall Officials: Eric Swanson, M.D., Principal Investigator — Swanson Cener
Locations (1):
- Swanson Center, Leawood, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Comerota AJ, Chouhan V, Harada RN, Sun L, Hosking J, Veermansunemi R, Comerota AJ Jr, Schlappy D, Rao AK. The fibrinolytic effects of intermittent pneumatic compression: mechanism of enhanced fibrinolysis. Ann Surg. 1997 Sep;226(3):306-13; discussion 313-4. doi: 10.1097/00000658-199709000-00010. PMID 9339937
- [Background] Swanson E. Do Sequential Compression Devices Really Reduce the Risk of Venous Thromboembolism in Plastic Surgery Patients? Plast Reconstr Surg. 2015 Oct;136(4):577e-578e. doi: 10.1097/PRS.0000000000001587. No abstract available. PMID 26114974
- [Background] Murphy RX Jr, Alderman A, Gutowski K, Kerrigan C, Rosolowski K, Schechter L, Schmitz D, Wilkins E. Evidence-based practices for thromboembolism prevention: summary of the ASPS Venous Thromboembolism Task Force Report. Plast Reconstr Surg. 2012 Jul;130(1):168e-175e. doi: 10.1097/PRS.0b013e318254b4ee. PMID 22743901
- [Background] Swanson E. Ultrasound screening for deep venous thrombosis detection: a prospective evaluation of 200 plastic surgery outpatients. Plast Reconstr Surg Glob Open. 2015 Apr 7;3(3):e332. doi: 10.1097/GOX.0000000000000311. eCollection 2015 Mar. PMID 25878943